CLINICAL TRIAL: NCT07315750
Title: A Randomized Controlled Phase III Study to Evaluate the Combination of Disitamab Vedotin, Trastuzumab, and Tislelizumab Versus Chemotherapy (CAPOX) Combined With Trastuzumab With or Without Pembrolizumab as First-Line Treatment for Advanced Gastric/Gastroesophageal Junction Adenocarcinoma With HER2-high Expression
Brief Title: A Study of Disitamab Vedotin Combined With Trastuzumab and Tislelizumab Versus Chemotherapy Combined With Trastuzumab With or Without Pembrolizumab in HER2-high Expression Advanced Gastric or Gastroesophageal Junction Adenocarcinoma.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C040
Record Dates: First submitted 2025-12-03; First posted 2026-01-02 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Gastric Carcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — disitamab vedotin; tislelizumab; Oxaliplatin; Capecitabine; Trastuzumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Disitamab Vedotin Combined with Trastuzumab and Tislelizumab (Experimental): Participants will receive Disitamab Vedotin, Trastuzumab and Tislelizumab until the occurrence of intolerable toxicity, disease progression (investigator-assessed), initiation of new anti-tumor therapy, loss to follow-up, withdrawal of informed consent, or death (whichever occurs first).
  Interventions: Drug: Disitamab Vedotin; Drug: Tislelizumab; Drug: Trastuzumab
- Chemotherapy (CAPOX) Combined with Trastuzumab With or Without Pembrolizumab (Active Comparator): Participants will receive CAPOX, Trastuzumab and Trastuzumab. Only subjects whose PD-L1 expression is confirmed as CPS ≥1 by the central laboratory will receive pembrolizumab. Treatment will continue until the occurrence of intolerable toxicity, disease progression (investigator-assessed), initiation of new anti-tumor therapy, loss to follow-up, withdrawal of informed consent, or death (whichever occurs first).
  Interventions: Drug: CAPOX (oxaliplatin/capecitabine); Drug: Trastuzumab; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Disitamab Vedotin — Disitamab Vedotin: 2.5 mg/kg, IV, D1, Q2W;
  Arms: Disitamab Vedotin Combined with Trastuzumab and Tislelizumab
Drug: Tislelizumab — Tislelizumab: 200 mg, IV, D1, Q3W
  Arms: Disitamab Vedotin Combined with Trastuzumab and Tislelizumab
Drug: CAPOX (oxaliplatin/capecitabine) — Oxaliplatin: 130 mg/m², IV, D1, Q3W; Capecitabine: 1000 mg/m², po, BID, D1-D14, Q3W;
  Arms: Chemotherapy (CAPOX) Combined with Trastuzumab With or Without Pembrolizumab
Drug: Trastuzumab — Trastuzumab: Initial dose of 8mg/kg, followed by 6 mg/kg, IV, D1, Q3W;
Drug: Pembrolizumab — Pembrolizumab: 200mg, IV, D1, Q3W
  Arms: Chemotherapy (CAPOX) Combined with Trastuzumab With or Without Pembrolizumab

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Disitamab Vedotin combined with Trastuzumab and Tislelizumab Versus Chemotherapy Combined with Trastuzumab with or without Pembrolizumab as First-Line Treatment for Advanced Gastric/Gastroesophageal Junction Adenocarcinoma with HER2-high Expression.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily consent to participate in the study and sign the informed consent form
* Expected survival period >12 weeks
* ECOG Performance Status 0 or 1
* Histologically confirmed unresectable locally advanced or metastatic --gastric/gastroesophageal junction adenocarcinoma
* No prior systemic therapy for locally advanced or metastatic gastric cancer; or disease progression or recurrence occurring ≥6 months after completion of neoadjuvant/adjuvant therapy
* HER2-high expression
* At least one assessable lesion according to RECIST v1.1 criteria
* Adequate organ function
* Female subjects of childbearing potential must have a negative blood pregnancy test within 7 days prior to the first treatment, and agree not to breastfeed or donate ova from the signing of the informed consent form until 6 months after the last treatment. Male subjects must agree not to donate sperm from the signing of the informed consent form until 6 months after the last treatment.
* Able to understand the study requirements and willing to comply with the study and follow-up procedures

Exclusion Criteria:

* Presence of central nervous system (CNS) metastasis and/or carcinomatous meningitis
* Peripheral neuropathy > Grade 1
* Tumor lesions with a tendency to bleed
* Severe gastrointestinal dysfunction that may affect drug intake, transport, or absorption
* Bone metastases with a risk of paraplegia
* Past or current interstitial lung disease, or severely impaired lung function
* Other malignancies within 5 years prior to randomization, except for those expected to be cured with treatment
* Pregnant or breastfeeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 555 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (assessed by the BIRC) | 24 months
  Progression-free survival (PFS) is defined as the time from the date of randomization to disease progression per RECIST 1.1 as assessed by Blinded Independent Review Committee (BIRC) or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival | up to 5 years
  Overall survival (OS) refers to the time from the date of randomization to the date of death from any cause.
Progression-Free Survival (assessed by the investigator) | 24 months
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 as assessed by investigators or death due to any cause, whichever occurs first.
Objective Response Rate (assessed by the BIRC and investigators) | 24 months
  ORR is defined as the percentage of subjects who have a Complete Response (CR) or Partial Response (PR) per RECIST 1.1 as assessed by BICR and investigators .
Disease Control Rate (assessed by the BIRC and investigators) | 24 months
  DCR is defined as the proportion of subjects whose BOR is rated as CR, PR, or stable disease (SD) per RECIST 1.1 as assessed by BICR/ investigators .
Duration of Response (assessed by the BIRC and investigators) | 24 months
  For participants who demonstrate CR or PR, DOR is defined as the time from first response (CR or PR) to subsequent disease progression or death from any cause, whichever occurs first.
Patient-Reported Outcomes (EORTC-QLQ-C30) | 24 months
  The EORTC-QLQ-C30 is a 30-item cancer-specific instrument consisting of 5 functional scales (physical, role, emotional, social and cognitive), 9 symptom scales/items (fatigue, nausea/vomiting, general pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties) and a global health status scale. Most items are scored 1 ("not at all") to 4 ("very much") except for the items contributing to the global health status/QoL, which are scored 1 ("very poor") to 7 ("excellent"). All raw domain scores are linearly transformed to a 0-100 scale with higher scores on symptoms indicate a worse health state.
Patient-Reported Outcomes (EORTCQLQ-STO22) | 24 months
  Quality of life in patients with colorectal cancer is assessed using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) STO22. It will be evaluated at Screening and Tumor Assessment Visit. The higher score means the worse quality of life.
Patient-Reported Outcomes (EQ-5D-5L) | 24 months
  EQ-5D-5L is a standardized instrument for use as a measure of health outcomes consisting of 6 items that cover 5 main domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and a general visual analog scale for health status.It was developed by the EuroQol Group for use as a generic, preference-based measure of health outcomes. Each dimension comprises 5 levels (no problems, slight problems, moderate problems, severe problems, extreme problems). A unique EQ-5D-5L health state is defined by combining 1 level from each of the 5 dimensions. This questionnaire also records the respondent's self-rated health status on a vertical graduated (0 = the worst health a participant can imagine to 100 = the best health a participant can imagine) visual analogue scale. Responses to the 5 items will also be converted to a weighted health state index (utility score) based on values derived from general population samples.
Adverse Events | 24 months
  Incidence, severity, and relationship to the investigational product of adverse events (AEs) and serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, BJ-Beijing, China